CLINICAL TRIAL: NCT00815048
Title: Remifentanil and Atropine for Intubation in Neonates; a Randomized Controlled Trial
Brief Title: Remifentanil and Atropine for Intubation in Neonates
Acronym: RAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: McMaster University (Other)
Responsible Party: Khalid AlFaleh, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RAIN
Record Dates: First submitted 2008-12-24; First posted 2008-12-29 (Estimated); Last update posted 2008-12-29 (Estimated); Status verified 2008-12

CONDITIONS: Endotracheal Intubation
Keywords: Remifentanil; Endotracheal intubation; Premedication; Sedation; Endotracheal Intubation in Neonates
MeSH Terms: interventions — Atropine; Remifentanil; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remifentanil (Active Comparator): Atropine
  Remifentanil
  Interventions: Drug: Atropine/Remifentanil
- Fentanyl (Placebo Comparator): Atropine
  Fentanyl
  Succinylcholine
  Interventions: Drug: Fentanyl/Atropine/Succinylcholine

INTERVENTIONS:
Drug: Atropine/Remifentanil — Atropine 20mcg/kg
  Remifentanil 3mcg/kg
  Arms: Remifentanil
Drug: Fentanyl/Atropine/Succinylcholine — Atropine 20mcg/kg
  Fentanyl 2mcg/kg
  Succinylcholine 2mg/kg
  Arms: Fentanyl

SUMMARY:
The investigators hypothesize that the use of a combination of Atropine and Remifentanil will safely facilitate non emergent intubation procedure as effectively as the protocol of Atropine, Fentanyl, and Succinylcholine.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable neonates of any gestational age admitted to the Neonatal Intensive Care Unit at McMaster Children's Hospital requiring an elective endotracheal intubation was anticipated.

Exclusion Criteria:

* Urgent intubations
* Cyanotic congenital heart lesions
* Anticipated difficult airway
* Concurrent or recently administered (within 3 hours of the procedure) intravenous opioid infusions
* Pre-existing hyperkalemia
* Family history of malignant hyperthermia
* Prior enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Time to Successful intubation | 15 minutes

SECONDARY OUTCOMES:
Time to return of spontaneous respirations | 15 minutes
Oxygen saturation | During the procedure up to 15 minutes
Heart Rate | During the procedure up to 15 minutes
Blood Pressure | During the procedure up to 15 minutes
Intubation Condition | 15 minutes post procedure
Evidence of Trauma | 15 minutes post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Khalid M Alfaleh, MBBS, MSc, Principal Investigator — King Saud University; Karen Choong, FRCPC, Study Director — McMaster University
Locations (1):
- McMaster University NICU, Hamilton, Ontario, Canada